CLINICAL TRIAL: NCT03314740
Title: Italian Multicenter Randomized Phase II Study of Weekly Paclitaxel vs. Cediranib-Olaparib (Continuous vs. Intermittent) in Patients With Platinum Resistant High Grade Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Best Approach in Recurrent-Ovarian-Cancer-with Cediranib-Olaparib
Acronym: BAROCCO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRFMN-OVA-7289
Record Dates: First submitted 2017-06-01; First posted 2017-10-19 (Actual); Results first posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Drug Therapy; cediranib; Tyrosine Kinase Inhibitors; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Active Comparator): Intravenous administration of weekly Paclitaxel (dosage: 80 mg/mq) for a maximum of 6 cycles. Cycle is defined as 4 weeks.
  Interventions: Drug: Paclitaxel
- Arm B (Experimental): Oral administration of two experimental drugs:
  * Cediranib 20 mg/day given 7 days per week
  * Olaparib 600 mg / day (i.e. 300 mg twice a day) 7 days per week until progression, unacceptable toxicity, patient or physician decision to discontinue or death.
  Interventions: Drug: Cediranib; Drug: Olaparib
- Arm C (Experimental): Oral administration of two experimental drugs:
  * Cediranib 20 mg/day given 5 days per week
  * Olaparib 600 mg / day (i.e. 300 mg twice a day) 7 days per week until progression, unacceptable toxicity, patient or physician decision to discontinue or death.
  Interventions: Drug: Cediranib; Drug: Olaparib

INTERVENTIONS:
Drug: Paclitaxel — Comparator active compound
  Other Names: chemotherapy
  Arms: Arm A
Drug: Cediranib — Experimental compound
  Other Names: tyrosine kinase inhibitor
  Arms: Arm B; Arm C
Drug: Olaparib — Experimental compound
  Other Names: Parp inihibitor
  Arms: Arm B; Arm C

SUMMARY:
This is a Phase II, randomized, multi-centre study aiming at comparing the efficacy of Olaparib and Cediranib vs. weekly Paclitaxel in terms of progression free survival (PFS) in platinum refractory or resistant recurrent ovarian cancer.

Patients will be randomised in a 1:1:1 ratio to three treatment arms:

* Arm A: Paclitaxel 80 mg/mq every week
* Arm B: Cediranib 20 mg/day + Olaparib 600 mg / day (i.e. 300 mg BD) given every day
* Arm C: Cediranib 20 mg/day given 5 days per weeks + Olaparib 600 mg / day (i.e. 300 mg BD) given 7 days per weeks

DETAILED DESCRIPTION:
Both the experimental arms (Arm B and C) will be compared with Arm A in terms of PFS.

If both superior to the control (Arm A), they will be compared in terms of gastrointestinal safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients affected by pathologically confirmed high-grade epithelial ovarian, fallopian tube, or primary peritoneal cancer.
2. Relapsed/progressive disease within 6 months from last platinum-based chemotherapy (platinum resistant/refractory disease).
3. Any line of treatment (after the first).
4. Any "last" chemotherapy line, including Paclitaxel, that should have been administered at least 6 months before the study beginning.
5. Patients must be women > 18 years of age.
6. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

   * Haemoglobin ≥ 10.0 g/dL and no blood transfusions in the 28 days prior to entry/randomization - Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * White blood cells (WBC) > 3x109/L
   * Platelet count ≥ 100 x 109/L
   * Total bilirubin ≤ 1.5 x institutional Upper Limit of Normal (ULN)
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional Upper Limit of Normal, unless liver metastases are present in which case it must be ≤ 5x ULN
   * Creatinine clearance estimated using the Cockcroft-Gault equation ≥51 mL/min,.
7. ECOG performance status 0-1.
8. Patients must have a life expectancy ≥ 16 weeks.
9. Evidence of non-childbearing status for women of childbearing potential (negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1 or postmenopausal women. Postmenopausal status is defined as:

   * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
   * LH and FSH levels in the post-menopausal range for women under 50
   * Radiation-induced oophorectomy with last menses >1 year ago,
   * Chemotherapy-induced menopause with >1 year interval since last menses
   * Surgical sterilization (bilateral oophorectomy or hysterectomy)
10. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment, scheduled visits and examinations including follow up.
11. At least one lesion (measurable as defined by RECIST 1.1) that can be accurately assessed by CT scan or MRI with Chest X-ray at baseline and follow up visits.
12. BRCA1-2 mutation status known. In case of BRCA status unknown, the BRCA test must be performed before the randomization or, if not feasible, within the end-of the study treatment.
13. Provision of informed consent prior to any study specific procedures. In case of patients unable to give written informed consent, is necessary to have the subject or legal representative sign, but in any case a witness must be present and sign and date with the person providing informed consent.

Exclusion Criteria:

1. Any previous treatment with a PARP inhibitor, including Olaparib.
2. Prior treatment with Cediranib (previous bevacizumab or other antiangiogenic drugs are allowed)
3. Previous progression to weekly Paclitaxel
4. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years
5. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive bisphosphonates for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment with study drug.
6. Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting Olaparib is 2 weeks.
7. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting Olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
8. Persistent toxicities (>=CTCAE grade 2) with the exception of alopecia, caused by previous cancer therapy.
9. Resting ECG with QTc > 470msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
10. Greater than +1 proteinuria on two consecutive dipsticks taken no less than 1 week apart unless urinary protein < 1.5g in a 24 hr period or urine protein/creatinine ratio < 1.5.
11. A history of poorly controlled hypertension or resting blood pressure >150/100 mmHg in the presence or absence of a stable regimen of anti-hypertensive therapy (measurements will be made after the patient has been resting supine for a minimum of 5 minutes. Two or more readings should be taken at 2-minute intervals and averaged. If the first two diastolic readings differ by more than 5 mmHg, then an additional reading should be obtained and averaged).
12. Blood transfusions within 28 days prior to study start.
13. Features suggestive of Myelodysplastic syndrome or Acute myeloid leukemia (MDS/AML) on peripheral blood smear.
14. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 28 days prior to treatment.
15. Major surgery within 4 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
16. Patients considered at poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, unstable spinal cord compression (untreated and unstable for at least 28 days prior to study entry), superior vena cava syndrome, extensive bilateral lung disease on HRCT scan or any psychiatric disorder that prohibits obtaining informed consent.
17. Patients unable to swallow medications and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
18. Breast feeding women.
19. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV) and are receiving antiviral therapy.
20. Patients with known active hepatic disease (i.e., Hepatitis B or C).
21. Patients with a known hypersensitivity to Olaparib, Cediranib or any of the excipients of the products.
22. Patients with a known hypersensitivity to Paclitaxel.
23. Patients with uncontrolled seizures.
24. History of abdominal fistula or gastrointestinal perforation.
25. Prior gastrectomy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients affected by uro-genital neoplasm of ovary.
Enrollment: 123 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roldano Fossati, MD, Study Director — Mario Negri Institute for Pharmacological Research; Nicoletta Colombo, MD, Principal Investigator — European Institute of Oncology
Locations (6):
- Italy (6):
  - Spedali Civili di Brescia, Brescia, BS
  - Ospedale San Gerardo - ASST Monza, Monza, MB
  - Istituto Oncologico Veneto (IOV), Padua, PD
  - Arcispedale Santa Maria Nuova, Reggio Emilia, RE
  - Policlinico Umberto I - Università La Sapienza, Rome, RM
  - Istituto Eurpeo di Oncologia (IEO), Milan

REFERENCES:
- [Derived] Tattersall A, Ryan N, Wiggans AJ, Rogozinska E, Morrison J. Poly(ADP-ribose) polymerase (PARP) inhibitors for the treatment of ovarian cancer. Cochrane Database Syst Rev. 2022 Feb 16;2(2):CD007929. doi: 10.1002/14651858.CD007929.pub4. PMID 35170751
- [Derived] Colombo N, Tomao F, Benedetti Panici P, Nicoletto MO, Tognon G, Bologna A, Lissoni AA, DeCensi A, Lapresa M, Mancari R, Palaia I, Tasca G, Tettamanzi F, Alvisi MF, Rulli E, Poli D, Carlucci L, Torri V, Fossati R, Biagioli E; BAROCCO study group. Randomized phase II trial of weekly paclitaxel vs. cediranib-olaparib (continuous or intermittent schedule) in platinum-resistant high-grade epithelial ovarian cancer. Gynecol Oncol. 2022 Mar;164(3):505-513. doi: 10.1016/j.ygyno.2022.01.015. Epub 2022 Jan 19. PMID 35063281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was approved and activated in 7 experimental sites. The enrolment was closed on 18th October 2018 with the inclusion of 123 patients.
Groups:
- Arm B: Oral administration of two experimental drugs:
  * Cediranib 20 mg/day given 7 days per week
  * Olaparib 600 mg / day (i.e. 300 mg twice a day) 7 days per week until progression, unacceptable toxicity, patient or physician decision to discontinue or death.
  Cediranib: Experimental compound
  Olaparib: Experimental compound
- Arm C: Oral administration of two experimental drugs:
  * Cediranib 20 mg/day given 5 days per week
  * Olaparib 600 mg / day (i.e. 300 mg twice a day) 7 days per week until progression, unacceptable toxicity, patient or physician decision to discontinue or death.
  Cediranib: Experimental compound
  Olaparib: Experimental compound
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C
Started | 41 | 41 | 41
Completed | 41 | 41 | 41
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Total
Number analyzed (Participants) | 41 | 41 | 41 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (8.1) | 61.0 (11.4) | 61.4 (9.4) | 61.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 41 | 123
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 36 | 38 | 40 | 114
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 0 | 6
Previous Chemotherapy lines [Mean (Standard Deviation); unit: lines] — Chemotherapy treatments received before the study entry
  lines | 2.6 (1.2) | 3.1 (1.5) | 2.9 (1.2) | 2.9 (1.3)
BRCA mutated [Count of Participants; unit: Participants] — Blood test for BRCA1-2 germline mutations. If one of the two genes resultes as mutated the patient is considered as BRCA mutated
  Participants | 4 | 7 | 4 | 15
Last Platinum Free interval [Mean (Standard Deviation); unit: months] — Time interval between the day of the last platinum treatment administration and the last progression
  months | 3.0 (2.3) | 2.5 (1.9) | 2.3 (2.4) | 2.6 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Progression Free Survival (PFS)
Description: PFS is defined as time from randomization to the date of first progression or death for any cause, whichever comes first.
  Progression was established as the radiological disease progression according to RECIST 1.1 (as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions") or to clinical assessment in case radiological evaluation is not feasible due to clinical condition.
Time Frame: An average of 30 months for each participant
Population: Intention to treat population
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 41 | 41 | 41
months | 3.1 [1.9 to 6.3] | 5.6 [3.2 to 7.4] | 3.8 [2.0 to 5.8]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; p = 0.265, cox model; Hazard Ratio (HR) = 0.76, 90% CI 2-sided [0.5 to 1.14]
Statistical Analysis 2: Comparison: Arm A vs Arm C; Test type: Superiority; p = 0.904, cox- model; Hazard Ratio (HR) = 1.03, 90% CI 2-sided [0.68 to 1.55]

2. Primary Outcome: Safety: Number of Evacuations Per Day
Description: Number of evacuations per day used as an index of gastro-intestinal toxicity profile of experimental drugs
Time Frame: Evacuation were collected daily for the first four weeks of treatment of experimental drugs
Population: No primary safety analysis in terms of gastrointestinal events between continuous and intermittent arm was done because neither experimental arm showed any superiority in PFS over the control arm.
Arm/Group | Arm B | Arm C
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Efficacy: Objective Response Rate (ORR)
Description: Percentage of patients with an objective response as determined by RECIST 1.1
Time Frame: Disease assessments were scheduled every 8 weeks (+/- 1 week) from randomization for all treatment duration (an average of 3.5 months).
Population: ORR population: patients in the ITT population who received at least one dose of study treatment and had at least one radiological assessment.
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 24 | 39 | 36
participants | 9 | 6 | 4

4. Secondary Outcome: Efficacy: PFS2
Description: PFS2 is defined as time from first progression to the date of second progression or death for any cause, whichever comes first.
Time Frame: Up to one year after the last patient enrolled
Reporting Status: Not Posted

5. Secondary Outcome: Efficacy: Overall Survival (OS)
Description: OS is defined as time from randomization to the date of death for any cause
Time Frame: Up to one year after the last patient enrolled
Reporting Status: Not Posted

6. Secondary Outcome: Efficacy: Quality of Life
Description: Quality of Life evaluated by the Functional Assessment of Cancer Therapy-Ovarian (FACT-O) questionnaire
Time Frame: Up to sixth month of study treatment
Reporting Status: Not Posted

7. Secondary Outcome: Safety: Maximum Toxicity Grade
Description: Maximum toxicity grade experienced by each patient, for each toxicity, according to NCI-CTCAE v. 4.03
Time Frame: Up to 30 days after the end of treatment
Reporting Status: Not Posted

8. Secondary Outcome: Safety: Number of Patients Experiencing Grade 3-4 Toxicity for Each Toxicity
Description: Number of patients experiencing grade 3-4 toxicity for each toxicity according to NCI-CTCAE v. 4.03
Time Frame: Adverse events were collected at the end of each cycle for the duration of treatment for each participant (an average of 3.5 months) and following 30 days after the end of treatment.
Population: safety population: randomized patients receiving at least one dose of study drugs
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 28 | 41 | 41
Participants
  Anemia grade≥3 | 0 | 4 | 6
  Bone marrow hypocellular grade≥3 | 0 | 1 | 0
  Febrile neutropenia grade≥3 | 0 | 0 | 1
  Diarrhea grade≥3 | 0 | 2 | 1
  Mucositis oral grade≥3 | 0 | 1 | 0
  Nausea grade≥3 | 0 | 1 | 3
  Vomiting grade≥3 | 0 | 0 | 2
  Fatigue grade≥3 | 0 | 4 | 5
  Sepsis grade 5 | 1 | 0 | 0
  Neutrophil count decreased grade≥3 | 2 | 1 | 1
  Platelet count decreased grade≥3 | 0 | 1 | 0
  White blood cells decreased grade≥3 | 1 | 0 | 0
  Anorexia grade≥3 | 0 | 1 | 0
  Myelodysplastic syndrome grade 5 | 0 | 1 | 0
  Peripheral motor neuropathy grade≥3 | 1 | 0 | 0
  Pneumonitis grade≥3 | 0 | 1 | 0
  Palmar-plantar erythrodysesthesia syndrome grade≥3 | 0 | 1 | 0
  Hypertension grade≥3 | 0 | 5 | 6
  Thromboembolic event grade≥3 | 0 | 0 | 1

9. Secondary Outcome: Safety: Type, Frequency and Nature of SAEs
Description: Type, frequency and nature of SAEs, according to NCI-CTCAE v. 4.03
Time Frame: Up to 30 days after the end of treatment
Reporting Status: Not Posted

10. Secondary Outcome: Safety: Number of Patients With at Least a SAE; Patients With at Least a SADR
Description: Number of patients with at least a SAE; patients with at least a SADR, according to NCI-CTCAE v. 4.03
Time Frame: Up to 30 days after the end of treatment
Reporting Status: Not Posted

11. Secondary Outcome: Safety: Number of Patients With at Least a SUSAR
Description: Number of patients with at least a SUSAR, according to NCI-CTCAE v. 4.03
Time Frame: Up to 30 days after the end of treatment
Reporting Status: Not Posted

12. Secondary Outcome: Compliance: Number of Administered Cycles
Description: The endpoint for compliance is the number of administered cycles.
Time Frame: Up to one year after the last patient enrolled
Reporting Status: Not Posted

13. Secondary Outcome: Compliance: Reasons for Discontinuation and Treatment Modification
Description: The endpoints for compliance are the reasons for discontinuation and treatment modification.
Time Frame: Up to one year after the last patient enrolled
Reporting Status: Not Posted

14. Secondary Outcome: Compliance: Dose Intensity
Description: Entire dose administered during treatment
Time Frame: Up to one year after the last patient enrolled
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected at the end of each cycle for the duration of treatment for each participant (an average of 3.5 months) and following 30 days after the end of treatment.
Description: Only patients receiving at least one dose of treatment were analysed
Arm/Group | Arm A | Arm B | Arm C
All-Cause Mortality (participants affected / at risk) | 24/28 | 31/41 | 34/41
Serious Adverse Events (participants affected / at risk) | 3/28 | 11/41 | 9/41
Other Adverse Events (participants affected / at risk) | 16/28 | 36/41 | 34/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=28) | Arm B (N=41) | Arm C (N=41)
abdomina pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (3) | 5 (5)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=28) | Arm B (N=41) | Arm C (N=41)
Anemia (Blood and lymphatic system disorders) | 9 (14) | 6 (20) | 9 (16)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 6 (22) | 3 (5)
Nausea (Gastrointestinal disorders) | 6 (8) | 24 (39) | 22 (33)
Vomiting (Gastrointestinal disorders) | 1 (1) | 18 (36) | 17 (27)
Fatigue (General disorders) | 9 (16) | 21 (41) | 17 (29)
Neutrophil count decreased (Investigations) | 3 (16) | 3 (5) | 2 (5)
Hypertension (Vascular disorders) | 1 (1) | 13 (21) | 9 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT03314740/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT03314740/SAP_001.pdf